CLINICAL TRIAL: NCT05655455
Title: The Effects of Dance and Movement Therapy Techniques and Walking Interventions on the Levels of Loneliness and Self-neglect in Elderly Aged 65 Years and Over
Brief Title: Dance and Movement Therapy Techniques in Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Gozde Yıldız Daş Geçim, assist.prof., Amasya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AmasyaU10
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Dance Therapy; Self Neglect; Loneliness
Keywords: old age; elderly; elder self neglect; level of loneliness

STUDY DESIGN:
Intervention Model Description: A repeated-measurement and 3-arm randomized controlled trial with pretest-posttest control group
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- experimental group 1 (Experimental): group 1: walking group
  Interventions: Behavioral: walking group: 1.group
- experimental group 2 (Experimental): group 2: dance and movement therapy group
  Interventions: Behavioral: dance and movement therapy group: 2.group
- control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: walking group: 1.group — In the study, walking attempt will be applied (2 x40 min/week and 6 weeks in total) to the 1st intervention group (n:15) in a gym. It will be given by a specialist in public health nursing. (first researcher)
  Arms: experimental group 1
Behavioral: dance and movement therapy group: 2.group — In the study, dance and movement therapy will be applied (2 x40 min/week and 6 weeks in total) to the 2nd intervention group (n:15) in a gym. It will be given by a specialist in psychiatric nursing.
  Arms: experimental group 2

SUMMARY:
Aim: To investigate the effects of dance and movement therapy or walking interventions for elderly people aged 65 and over who are registered to the family health center located in the city center of Amasya, on the loneliness and self-neglect levels of the elderly.

Method: In this study, which is a repeated-measurement and 3-armed randomized controlled study with a pretest-posttest control group, the elderly aged 65 and over will be randomly assigned to two 15-person experiments and a control group. In the study, dance and movement therapy techniques will be applied to the 1st intervention group (n:15), and walking attempt (2 x40 min/week and 6 weeks in total) to the 2nd intervention group (n:15). The data collection tool will be applied before the intervention and at the 1st and 3rd months after the intervention.

Conclusion: The main result of the study is to determine that dance and movement therapy and walking attempts for the elderly are effective in reducing the levels of loneliness and self-neglect in the elderly. It is thought that the results of the study will support the elderly mentally, socially and culturally and will guide the programs that will improve the health of the elderly.

DETAILED DESCRIPTION:
Introduction: The feeling of loneliness and self-neglect, which can be seen in all age groups and is an uncomfortable situation for individuals, are important factors that affect the physical and mental health and quality of life of individuals, which are more common in older ages. Coping with emotional, physical and social support networks to cope with the factors that cause the feeling of loneliness in the elderly, and applying programs that address all the variables that will prevent the decrease in the life satisfaction of the elderly as a result of loneliness reduce the feeling of self-neglect and loneliness in the elderly.

Aim: To investigate the effects of dance and movement therapy or walking interventions for elderly people aged 65 and over who are registered to the family health center located in the city center of Amasya, on the loneliness and self-neglect levels of the elderly.

Method: In this study, which is a repeated-measurement and 3-armed randomized controlled study with a pretest-posttest control group, the elderly aged 65 and over will be randomly assigned to two 15-person experiments and a control group. In the study, dance and movement therapy techniques will be applied to the 1st intervention group (n:15), and walking attempt (2 x40 min/week and 6 weeks in total) to the 2nd intervention group (n:15). The data collection tool will be applied before the intervention and at the 1st and 3rd months after the intervention.

Conclusion: The main result of the study is to determine that dance and movement therapy and walking attempts for the elderly are effective in reducing the levels of loneliness and self-neglect in the elderly. It is thought that the results of the study will support the elderly mentally, socially and culturally and will guide the programs that will improve the health of the elderly.

ELIGIBILITY:
Inclusion Criteria:

*65 years and older,

* Having no vision and hearing problems,
* Diagnosed and not having a chronic disease that would prevent participation in the study,
* Not having a diagnosed mental health problem,
* Does not have a disease that prevents physical exercise,

Exclusion Criteria:

* have a known physical or neurological disease

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
loneliness scale for elderly | 6 months
  Loneliness is one of the primary outcomes. This will be measured using the 'Loneliness Level Scale for the Elderly' scale. This scale is scored between 0-22; higher scores shows higher level of loneliness.
Elder Self-Neglect Scale | 6 months
  Self-neglect is the other primary outcome for this study. This will be measured using the 'Self-Neglect Scale in the Elderly' scale. This scale is scored between 60-300; higher scores shows higher level of self-neglect.

CONTACTS AND LOCATIONS:
Overall Officials: gozde yildiz das gecim, PhD, Principal Investigator — Amasya University
Locations (1):
- Amasya University Faculty of Health Sciences, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No